CLINICAL TRIAL: NCT03777813
Title: Association of Radiochemotherapy and Immunotherapy for the Treatment of Unresectable Oesophageal caNcer: a Comparative Randomized Phase II Trial
Brief Title: Association of Radiochemotherapy and Immunotherapy for the Treatment of Unresectable Oesophageal caNcer
Acronym: ARION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-110/1719 -PRODIGE 67-UCGI33; 2018-000708-40 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-09

CONDITIONS: Esophagus Cancer; Unresectable Malignant Neoplasm
Keywords: oesophagus; localised unresectable; adenocarcinoma or squamous cell carcinoma; durvalumab; FOLFOX 4 simplified; Definitive modulated-intensity radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — durvalumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Concomitant administration of durvalumab (dose: 1500 mg):
  Every 4 weeks during concurrent FOLFOX and after FOLFOX completion (total of 12 months of treatment)
  Definitive modulated-intensity radiotherapy will be delivered according to boost integrated technique 5 days a week for 5 weeks at a dose of:
  * 50 Gy delivered in 25 fractions to the macroscopic disease (endoscopic, TDM and fused FDG PET)
  * 45 Gy to the adjacent peri tumoral mucosis and prophylactic lymph node
  FOLFOX 4 simplified protocol, 1 infusion every 2 weeks during 3 months starting with radiotherapy (+/- 1 day):
  * IV oxaliplatin 85 mg/m² in 2 h on D1
  * IV Leucovorin 200 mg/m² in 2 h on D1, followed by
  * IV 5-FU 400 mg/m² in 10 minutes on D1 followed by
  * IV continuous infusion 5-FU 2400 mg/m² in 46 h
  Interventions: Drug: Durvalumab; Combination Product: IMRT 50 Gy + FOLFOX4 simplifIed (oxaliplatin, leucovorin, 5-FU)
- Arm B (Active Comparator): Definitive modulated-intensity radiotherapy will be delivered according to boost integrated technique 5 days a week for 5 weeks at a dose of:
  * 50 Gy delivered in 25 fractions to the macroscopic disease (endoscopic, TDM and fused FDG PET)
  * 45 Gy to the adjacent peri tumoral mucosis and prophylactic lymph node
  FOLFOX 4 simplified protocol, 1 infusion every 2 weeks during 3 months starting with radiotherapy (+/- 1 day):
  * IV oxaliplatin 85 mg/m² in 2 h on D1
  * IV Leucovorin 200 mg/m² in 2 h on D1, followed by
  * IV 5-FU 400 mg/m² in 10 minutes on D1 followed by
  * IV continuous infusion 5-FU 2400 mg/m² in 46 h
  Interventions: Combination Product: IMRT 50 Gy + FOLFOX4 simplifIed (oxaliplatin, leucovorin, 5-FU)

INTERVENTIONS:
Drug: Durvalumab — Radiochemotherapy in standard arm and in experimental arm: 10 weeks (RT 50 Gy and FOLFOX q2w) Immunotherapy in experimental arm only: Patients will received concomitantly a maximum of 12 infusions
  Other Names: IMRT 50 Gy + FOLFOX4 simplifIed (oxaliplatin, leucovorin, 5-FU)
  Arms: Arm A
Combination Product: IMRT 50 Gy + FOLFOX4 simplifIed (oxaliplatin, leucovorin, 5-FU) — Radiochemotherapy in standard arm and in experimental arm: 10 weeks (RT 50 Gy and FOLFOX q2w)

SUMMARY:
This study aims to assess the efficacy of durvalumab in combination with radiochemotherapy (FOLFOX and IMRT) and then as maintenance therapy for treating patients with localised unresectable oesophageal cancer. This is a randomized, French national, multicentre, comparative phase II trial

DETAILED DESCRIPTION:
ARION study will randomize 120 patients, in 12 centers in France, according to a ratio 1:1 in the following arm of treatment:

- Standard and experimental arm:

Definitive modulated-intensity radiotherapy will be delivered according to boost integrated technique 5 days a week for 5 weeks at a dose of:

* 50 Gy delivered in 25 fractions to the macroscopic disease (endoscopic, TDM and fused FDG PET)
* 45 Gy to the adjacent peri tumoral mucosis and prophylactic lymph node

FOLFOX 4 simplified protocol, 1 infusion every 2 weeks (q2w) during 3 months starting with radiotherapy (+/- 1 day):

* IV oxaliplatin 85 mg/m² in 2 h on day 1 (D1)
* IV Leucovorin 200 mg/m² in 2 h on D1, followed by
* IV 5-FU 400 mg/m² in 10 minutes on D1 followed by
* IV continuous infusion 5-FU 2400 mg/m² in 46 h
* Experimental arm: Concomitant administration of durvalumab:

Every 4 weeks during concurrent FOLFOX (dose: 1500 mg) and after FOLFOX completion (total of 12 months of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous cell carcinoma or adenocarcinoma of the oesophagus,
2. Unresectable disease due to anatomical consideration or medical condition (patient unfit for surgical procedure),
3. Presence of at least one measurable lesion >10 mm with spiral CT scan,
4. No prior therapy for pathology investigated including chemotherapy or radiotherapy prior to the study, except anterior out of field radiotherapy, received for treatment of another primary tumor considered in remission, in the past 5 years,
5. Age ≥18 years old,
6. WHO performance status <2 (i.e., 0 or 1),
7. Body weight >35 kg,
8. Life expectancy of at least 12 weeks ,
9. Adequate haematology laboratory data within the 7 days before randomization

   1. Absolute neutrophils >1.5 x 109/L
   2. Platelets >100 x 109/L
   3. Haemoglobin ≥9 g/dL,
10. Adequate Biochemistry laboratory data within the 7 days before randomization

    1. Total bilirubin ≤1.5 x upper limit of normal (ULN)
    2. Transaminases ≤2.5 x ULN
    3. Alkaline phosphatases ≤5 x ULN,
    4. Measured creatinine clearance (CL) >40 mL/min by the Cockcroft-Gault formula,
    5. Glycaemia ≤1.5 x ULN
    6. Cholesterolaemia ≤7.30 mmol/L,
    7. Albumin >28 g/L
11. Adequate haemostasis laboratory data within 7 days prior to randomization: prothrombin time (PT) within the normal range,
12. Adequate values for calcium, potassium and magnesium levels measured within 7 days prior to randomization,
13. Women should be post-menopaused or willing to accept the use an effective contraceptive regimen during the treatment period and for at least 6 months after the end of the study. All non-menopausal women should have a negative pregnancy test within 72 h prior to randomization. Men should accept to use an effective contraception during treatment period and at least 6 months after the end of the study especially after the last dose of oxaliplatin treatment.
14. Patients must have provided consent for the study by signing and dating a written informed consent form prior to any study specific procedures, sampling, or analyses,
15. Patient affiliated to a social security regimen.
16. Uracilemia < 16ng/ml
17. Forced expiratory volume (FEV) >1 liter or > 50% of the theoretical value

Exclusion Criteria:

1. Previous treatment with another PD-1, PD-L1 including durvalumab or CTLA-4 inhibitor
2. Metastatic disease,
3. Patients should not receive live vaccine 30 days prior to study drug
4. Female patients who are pregnant or breastfeeding
5. Uncontrolled intercurrent illness including, but not limited to diabetes, hypertension, pulmonary failure, chronic renal or hepatic diseases, active peptic ulcer disease or gastritis, active bleeding, diatheses... (non-exhaustive list),
6. Clinically significant cardiac disease or impaired cardiac function, such as:

   1. Congestive heart failure requiring treatment (New York Heart Association [NYHA] grade ≥2), left ventricular ejection fraction (LVEF) <50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO), or uncontrolled arterial hypertension defined by blood pressure >140/100 mmHg at rest (average of 3 consecutive readings),
   2. History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, e.g. congenital long QT syndrome, high- grade/complete AV-blockage,
   3. Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), coronary angioplasty, or stenting), <3 months prior to screening,
   4. MeanQT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
7. Current or prior use of immunosuppressive medication within 28 days before the first administration of durvalumab (exception: systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or equivalent are allowed as well as steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) - Topical, inhaled, nasal, and ophthalmic steroids are allowed,
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stabilised with hormone replacement therapy
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with coeliac disease controlled by diet alone
9. Known primary immunodeficiency or active HIV,
10. Patient with a dihydropyrimidine dehydrogenase (DPD) deficiency (Uracilemia ≥ 16 ng/ml, the test should be done for all patients before 5-FU administration)* ,
11. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months indicated by positive HBS antibody test for hepatitis B or hepatitis C virus ribonucleic acid (HCV antibody),
12. History of organ transplantation requiring the use of immunosuppressive medication, including allogenic stem cell transplant
13. History of active tuberculosis or latent disease capable of reactivation,
14. Current pneumonitis or interstitial lung disease,
15. Other invasive malignancy within 2 years prior to entry into the study, except for those treated with surgical therapy only,
16. History of severe allergic reactions or hypersensitivity to any unknown allergens or any components of the study drug (refer to IB of durvalumab section 5.5.1.11).
17. Any prior corticosteroid-refractory immune-related adverse event (irAE),
18. Oeso-tracheal or oeso-bronchial fistulae,
19. Major surgery within 28 days prior to the first dose of study treatment
20. Toxicities of grade ≥1 from any previous therapy,
21. Peripheral sensory neuropathy with functional impairment
22. Severe infection requiring parenteral antibiotic treatment
23. Patients treated with sorivudine or analogues as brivudine
24. Patients treated with phenytoin for prophylaxis
25. Participation in another therapeutic trial within the 30 days prior to study inclusion,
26. Patients deprived of liberty or under guardianship,
27. Patients unable to adhere to the protocol for geographical, social, or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
cPFS (centrally reviewed cPFS) | 12-months cPFS
  defined by a blinded independent centralized revue of progression free survival. cPFS is defined as the time from randomization until progression or death; patients alive and without documented progression at last follow-up news have PFS censored at this date or at initiation of new anticancer treatment (if applicable). Progression will be defined with central external reviewing of TDM per RECIST v1.1

SECONDARY OUTCOMES:
Overall survival (OS) | For each treatment arms, survival rates (PFS and OS) will be estimated at 12, 18 and 24 months
  defined as the time between randomization and death due to any cause.
Adverse Events | 2 years after randomization
  will be assessed on occurrence of Adverse Events (AEs) based on NCI CTCAE v5.0
Quality of Life OES18, used for patients with oesophageal cancer always complemented by the QLQ-C30 measuring 5 functional scales (physical, everyday activity, cognitive, emotional and social) and 3 symptoms scales (fatigue, pain, nausea and vomiting) | 2 years after randomization
  scores EORTC QLQ C30 - OES18

CONTACTS AND LOCATIONS:
Overall Officials: Anouchka Modesto, Doctor, Principal Investigator — Institut Claudius Regaud; Laurent Quero, Doctor, Principal Investigator — Hôpital Saint Louis / Université Paris Diderot
Locations (7):
- France (7):
  - Centre Oscar Lambret, CLCC UNICANCER, Lille
  - Hôpital Saint Louis, APHP, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Universitaire, Poitiers
  - Centre Paul Strauss, CLCC UNICANCER, Strasbourg
  - Iuct, Clcc Unicancer, Toulouse
  - CHU Rangueil Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.